CLINICAL TRIAL: NCT01606722
Title: Relation Between Darunavir Levels and Virological Efficacy, Integrated Proviral ADN and Resistance Mutations in HIV-infected Patients on Treatment With Darunavir/Ritonavir Monotherapy
Brief Title: Darunavir Levels, Virological Efficacy, Proviral ADN and Resistances in Patients on Darunavir/Ritonavir Monotherapy
Acronym: MonDar
Status: Completed | Type: Observational
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Luis F. Lopez-Cortes, MD, PhD., Hospitales Universitarios Virgen del Rocío
Other Study IDs: LLC-DAR-2010-01; LLC-DAR-2010-01 (Other Grant/Funding Number: Consejeria de Salud. Junta de Andalucia (exp: PI-0448-2010))
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: HIV-infection
Keywords: Antiretroviral therapy; Boosted-Darunavir monotherapy; Resistance; Proviral DNA-HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (plasma and PBMC)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Darunavir-ritonavir monotherapy: HIV-infected patients with undetectable viral load for at least for 6 months on stable therapy and no darunavir related mutations in the HIV-protease gene
  Interventions: Drug: Darunavir/ritonavir

INTERVENTIONS:
Drug: Darunavir/ritonavir — Darunavir/ritonavir (800/100 mg once daily) monotherapy
  Other Names: Prezista/norvir

SUMMARY:
To evaluate the relationship between plasma and intracellular darunavir (DRV) concentrations and virological efficacy in HIV-infected patients on DRV/rtv monotherapy.

DETAILED DESCRIPTION:
To be enrolled, subjects had a plasma HIV-RNA <50 copies/mL for at least 6 months based, virologic failure while on a PI-containing regimen was allowed if the genotypic resistance tests showed no major resistance mutation associated to reduced susceptibility to DRV/rtv according to the International AIDS Society. Patients with transitory episodes of detectable plasma HIV-RNA viral load ("blip") preceded and followed by a plasma viral load <50 copies/mL without changes in antiretroviral treatment could also been included. The only exclusion criteria were pregnancy, hepatitis B coinfection and the concomitant use of drugs with potential major interactions with DRV/rtv pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years, starting an antiretroviral regimen based on darunavir-ritonavir (800/100 mg) once daily monotherapy between June 2010 and September 2010
* Plasma RNA-VIH < 50 copies/ml on stable antiretroviral treatment for ≥ 6 months
* Absence of resistance mutations in the protease gene, based on treatment history and/or genotypic resistance testing. that would decrease darunavir susceptibility

Exclusion Criteria:

* Pregnancy
* Chronic B hepatitis
* Genotypic resistance tests with evidence of resistance mutations in the protease gene that would decrease darunavir susceptibility
* Concomitant use of drugs with potentially adverse interactions with darunavir-ritonavir pharmacokinetics, such as rifampin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients who started an antiretroviral regimen based on darunavir-ritonavir (800/100 mg) once daily monotherapy between June 2010 and September 2010
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Virological efficacy | 48 and 96 weeks
  To correlate the plasma and intracellular (cell-associated)) DRV levels with the virological efficacy analyzed by the time to loss of virological response (TLOVR) algorithm, considering VF as either: 1) two consecutive viral load >200 copies/mL, 2) a unique HIV-RNA >200 copies/mL if followed by lost to follow-up, or 3) the reintroduction of nucleos(t)ides because any reason.

SECONDARY OUTCOMES:
Impact of viral breakthrough on DNA-HIV reservoirs and immunologic activation | 48 and 96 weeks
  Impact of blips and persistent viraemia on DNA-HIV reservoirs and immunologic activation

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Lopez-Cortes, MD, PhD., Study Chair — Hospital Universitario Virgen del Rocio. Sevilla. Spain
Locations (1):
- Hospital Universitarios Virgen del Rocio, Seville, Seville, Spain

REFERENCES:
- [Derived] Gutierrez-Valencia A, Torres-Cornejo A, BenMarzouk-Hidalgo OJ, Ruiz-Valderas R, Lluch A, Viciana P, Lopez-Cortes LF. Darunavir minimum plasma concentration and ritonavir-boosted darunavir monotherapy outcome in HIV-infected patients. Antivir Ther. 2014;19(5):443-7. doi: 10.3851/IMP2722. Epub 2014 Jan 16. PMID 24434370